CLINICAL TRIAL: NCT06974747
Title: Immunomodulatory Effect of Pleuran (β-glucan From Pleurotus Ostreatus) in Children With Recurrent Respiratory Tract Infections
Brief Title: Immunomodulatory Effect of Pleuran in Children With Recurrent Respiratory Tract Infections
Acronym: IPRRTI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pleuran, s.r.o. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IPRRTI
Record Dates: First submitted 2025-05-05; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Respiratory Tract Infection
Keywords: pleuran; beta-glucan; immunomodulation; prevention; respiratory tract infection; children
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active group (Experimental): Dietary supplement Imunoglukan P4H® chewable tablets (tablet containing IMG® 50 mg + Zinc 5 mg + Vitamin D 10 μg in 1 tablet)
  Dosage:
  up to 25 kg 1 tablet once daily for 3 months over 25 kg 2 tablets once daily for 3 months
  Interventions: Dietary Supplement: Imunoglukan P4H® chewable tablets
- Placebo group (Placebo Comparator): Active Placebo Comparator (tablet containing 5 mg zinc + 10 μg vitamin D3)
  Dosage:
  up to 25 kg 1 tablet once daily for 3 months over 25 kg 2 tablets once daily for 3 months
  Interventions: Dietary Supplement: Placebo chewable tablets

INTERVENTIONS:
Dietary Supplement: Imunoglukan P4H® chewable tablets — IMG® 50 mg + Zinc 5 mg + Vitamin D 10 μg in 1 tablet
  Arms: Active group
Dietary Supplement: Placebo chewable tablets — Zinc 5 mg + Vitamin D 10 μg in 1 tablet
  Arms: Placebo group

SUMMARY:
International, multicentre, prospective, randomized, double-blind, placebo-controlled study with a food supplement Imunoglukan P4H® chewable tablets to evaluate preventive effect on reduction of respiratory tract infections (RTIs) in children with a history of recurrent respiratory tract infections (RRTIs) in the previous infectious season prior enrolment.

Participants or their guardians will record the incidence and duration of RTIs in the Patient diary for 3 months.

DETAILED DESCRIPTION:
Study population:

Children aged 3-18 years with a history of RRTIs:

* Age 3 to 5 years (< 6 years): 6 or more upper or lower respiratory tract infections from October 2022 until the end of March 2023
* Age 6 to 18 years (≥ 6 years): 3 or more upper or lower respiratory tract infections from October 2022 until the end of March 2023

Study design:

International (Slovak republic, Czech republic, Serbia), multicentre (36), prospective, randomized, double-blind, placebo-controlled study

Primary endpoint:

To evaluate the effect of Imunoglukan P4H® chewable tablets (IMG®+ zinc+ vitamin D3) compared to the placebo group (zinc + vitamin D3) on:

• reduction in the number of RTIs episodes (total number)

Secondary endpoints:

To evaluate the effect of Imunoglukan P4H® chewable tablets (IMG®+ zinc+ vitamin D3) compared to the placebo group (zinc + vitamin D3) on:

* reduction in the number of episodes of RTI subtypes
* reduction in the duration of RTI episodes (total duration, RTI subtypes)
* reduction of the need for antibiotic (ATB) therapy
* reduction of the number of missed days at school/nursery due to RTI
* reduction of the number of missed working days due to RTIs
* reduction of the number of emergency department visits due to RTI
* reduction of the number of physician visits due to RTI
* tolerability and safety

Randomization:

* Active group: Imunoglukan P4H® chewable tablets (IMG® 50 mg + Zinc 5 mg + Vitamin D3 10 μg in 1 tablet):
* Placebo group: Placebo chewable tablets (Zinc 5 mg + Vitamin D 10 μg in 1 tablet) Dosage:
* up to 25 kg of body weight 1 tablet once a day for 3 months
* over 25 kg 2 tablets once a day for 3 months

Diagnostic procedures:

• Patient diary (Incidence and duration of RTIs)

ELIGIBILITY:
Inclusion criteria:

* signed informed consent
* age 3-18 years
* history of recurrent respiratory infections:

  * Age 3 to 5 years (< 6 years): 6 or more upper or lower respiratory tract infections from October 2022 until the end of March 2023
  * Ages 6 to 18 years (≥ 6 years): more than 3 upper or lower respiratory tract infections from October 2022 until the end of March 2023

Exclusion Criteria:

* refused informed consent
* bronchopulmonary dysplasia
* primary immunodeficiency
* cystic fibrosis
* chronic diarrhoea
* chronic diseases of the lungs, kidneys and liver
* malformations of the cardiovascular system
* oncological disease
* malnutrition
* intolerance to any of the ingredients in the study product
* taking preventive immunomodulatory therapy (beta-glucans, bacterial lysates, isoprinosine) less than 14 days prior enrolling the patient into the study

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 217 (Actual)
Dates: Start 2023-09-25 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
change in the number of RTIs episodes (total number) | change in the number of RTIs episodes (total number) during 3 month supplementation (from enrollment to the end of the treatment at 3 months)
  number of episodes of respiratory infections will be compared between the two study goups

SECONDARY OUTCOMES:
change in the number of episodes of RTI subtypes | change in the number of RTIs episodes (subtypes) during 3 month supplementation (from enrollment to the end of the treatment at 3 months)
change in the duration of RTI episodes (total duration, RTI subtypes) | change in the duration of RTIs episodes (total duration, subtypes) during 3 month supplementation (from enrollment to the end of the treatment at 3 months)
change in the number of antibiotic therapy courses | change in the number of antibiotic (ATB) therapy courses during 3 month supplementation (from enrollment to the end of the treatment at 3 months)
change of the number of missed days at school/nursery due to RTI | change of the number of missed days at school/nursery due to RTI during 3 month supplementation (from enrollment to the end of the treatment at 3 months)
change of the number of missed working days due to RTIs | change of the number of missed working days due to RTIs during 3 month supplementation (from enrollment to the end of the treatment at 3 months)
changeof the number of emergency department visits due to RTI | changeof the number of emergency department visits due to RTI during 3 month supplementation (from enrollment to the end of the treatment at 3 months)
change of the number of physician visits due to RTI | change of the number of physician visits due to RTI during 3 month supplementation (from enrollment to the end of the treatment at 3 months)
tolerability and safety | during 3 month supplementation (from enrollment to the end of the treatment at 3 months)
  monitoring the incidence of potential adverse events, incidence will be compared to placebo group

CONTACTS AND LOCATIONS:
Locations (3):
- IMUNOGLUKAN CZ, s.r.o., Prague, Czechia
- Medis Pharma d.o.o. Beograd, Belgrade, Serbia
- Imunoglukan, s.r.o., Bratislava, Slovakia

REFERENCES:
- [Derived] Jesenak M, Prokopova E, Bozensky J, Bonaci-Nikolic B, Milosevic K, Stankovic K, Ostojic O, Zivkovic Z, Diamant Z, Kunc P, Janeczek K, Majtan J. Novel Chewable Pleuran-Based Supplement Decreases Respiratory Tract Infections in Children: A Randomised Controlled Trial. Adv Ther. 2025 Dec;42(12):6132-6149. doi: 10.1007/s12325-025-03393-3. Epub 2025 Oct 14. PMID 41085920

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-06-30): https://cdn.clinicaltrials.gov/large-docs/47/NCT06974747/Prot_SAP_000.pdf
  • Informed Consent Form (2023-06-30): https://cdn.clinicaltrials.gov/large-docs/47/NCT06974747/ICF_001.pdf